CLINICAL TRIAL: NCT00149968
Title: Measurement of Patient Reported Gastrointestinal (GI) and Health-related Quality of Life (HRQL) Outcomes in Renal Transplant Recipients (MyLife)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ADE05
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2009-10

CONDITIONS: Renal Transplantation; Gastrointestinal Problems
Keywords: Renal transplantation; MMF; EC-MPS; GI problems
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myfortic (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS) — Patient on MMF treatment completes questionnaire and switch to equimolar doses of Myfortic. Maximum daily dose 1440 mg
  Other Names: Myfortic

SUMMARY:
The purpose of this study is to assess whether a switch from mycophenolate mofetil (MMF) to enteric-coated mycophenolate sodium (EC-MPS) results in improved GI- and/or health-related quality of life outcomes, and to determine the proportion of renal transplant recipients who are experiencing any GI complaints under MMF-based immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Received kidney transplant at least 3 months prior to study enrollment
* Receiving immunosuppressive regimen that includes MMF in combination with other immunosuppressive drugs
* Receiving MMF for at least 1 month prior to enrollment

Exclusion Criteria:

* Patients with any known hypersensitivity against mycophenolic acid, mycophenolate sodium, mycophenolate mofetil or other components of the formulations (e.g. lactose; see also summary of product characteristics of EC-MPS)
* If applicable, GI symptoms assumed or known not to be caused by MPA therapy (e.g. oral biphosphonates induced, infectious diarrhea)
* Acute rejection < 1 week prior to study enrollment

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Changes in gastrointestinal symptom severity after conversion from MMF to enteric-coated mycophenolate sodium | week 0, week 6-8

SECONDARY OUTCOMES:
Gastrointestinal symptoms under MMF-based immunosuppressive therapy | week 0, week 6-8
Assessment of quality of life, impact of immunosuppressive-induced gastrointestinal symptoms on patient's perception of symptom severity and quality of life | week 0, week 6-8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (2):
- Bonn, Germany
- Novartis, Basel, Switzerland

REFERENCES:
- [Background] Bolin P, Tanriover B, Zibari GB, Lynn ML, Pirsch JD, Chan L, Cooper M, Langone AJ, Tomlanovich SJ. Improvement in 3-month patient-reported gastrointestinal symptoms after conversion from mycophenolate mofetil to enteric-coated mycophenolate sodium in renal transplant patients. Transplantation. 2007 Dec 15;84(11):1443-51. doi: 10.1097/01.tp.0000290678.06523.95. PMID 18091520
- [Derived] Reinke P, Budde K, Hugo C, Petersen P, Schnuelle P, Fricke L, Scholz D, Sperschneider H, Bahner U, Kramer S, Fischer W, Arns W. Reduction of gastrointestinal complications in renal graft recipients after conversion from mycophenolate mofetil to enteric-coated mycophenolate sodium. Transplant Proc. 2011 Jun;43(5):1641-6. doi: 10.1016/j.transproceed.2011.01.184. PMID 21693250